CLINICAL TRIAL: NCT03453775
Title: Ultrasound-guided Lumbar Periradicular Injection: Effectiveness and Benefits of a Non Irradiating Infiltration Technique. A Randomized Controlled Trial
Brief Title: Ultrasound-guided Lumbar Periradicular Injection: a Non Irradiating Infiltration Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université Libre de Bruxelles (Other)
Responsible Party: Principal Investigator, Paul Gruson, Principal Investigator, Université Libre de Bruxelles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P2018/047
Record Dates: First submitted 2018-01-16; First posted 2018-03-05 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Low Back Pain; Sciatica; Disc, Herniated; Foraminal Hernia; Lumbar Foraminal Stenosis; Chronic Low Back Pain; Pain, Chronic; Injection Site Infiltration
MeSH Terms: conditions — Low Back Pain; Sciatica; Intervertebral Disc Displacement; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled, open trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound guided infiltration (Active Comparator): Ultrasound guided periradicular lumbar infiltration. Prone position. Lumbar spine level located in a median sagittal plane (spinous processes). High resolution curved 5MHz ultrasound probe. Probe is then rotated 90° for a median transverse image. Transverse plane translation towards desired side to have in the same plane: spinous process, vertebral blade, zygapophysial articulation, lateral facet, transverse process. Needle passes skin at 45° angle, directed "in plane" to the foramen. Fluoroscopy then performed to check needle's correct position. Poorly positioned needles will be replaced to obtain an intra-foraminal/epidural periradicular diffusion of the contrast medium. Once position is confirmed, Depomedrol 40mg + lidocaine 2% (1ml) is injected.
  Interventions: Device: Ultrasound guided periradicular lumbar infiltration
- Fluoroscopy guided infiltration (Active Comparator): Fluoroscopy guided periradicular lumbar infiltration. Prone position. Anatomical identification by radioscopy: antero-posterior and sagittal planes. Needle placement in an anteroposterior view, needle is then advanced in an inclined plane of 20° with respect to the initial axis, "tunnel vision" type image. Foramen is then reached in a sagittal view (not to progress too far in the intra-foraminal level). Needle progression is secured by neurostimulation (territory concerned by the root, intensity 0.2 milliampere to be at a distance of 1mm from the nerve root). Once needle is in place, fluoroscopy is performed to verify correct positioning (Omnipaque 300mg/ml of Iohexol, 0.2 to 0.5ml). Once position confirmed, mixture Depomedrol 40mg + lidocaine 2% (1ml) is injected.
  Interventions: Device: Fluoroscopy guided periradicular lumbar infiltration

INTERVENTIONS:
Device: Ultrasound guided periradicular lumbar infiltration — Once position of the needle is confirmed, the mixture Depomedrol 40mg + Lidocaine 2% (1ml) is injected, under neurostimulation with an intensity of 0.2 milliampere (identifies a distance of 1mm from the nerve root allowing the protection of the root of a lesion by the needle).
  Arms: Ultrasound guided infiltration
Device: Fluoroscopy guided periradicular lumbar infiltration — Once position of the needle is confirmed, the mixture Depomedrol 40mg + Lidocaine 2% (1ml) is injected, under neurostimulation with an intensity of 0.2 milliampere (identifies a distance of 1mm from the nerve root allowing the protection of the root of a lesion by the needle).
  Arms: Fluoroscopy guided infiltration

SUMMARY:
We propose here to evaluate the precision of lumbar periradicular infiltration performed under a transverse ultrasound approach by performing a fluoroscopic control once the needle in the desired position. The effectiveness of the technique will be assessed by measuring different pain and disability scores at four weeks post-infiltration: the Visual analogue pain Scale score, the DN4 score, and the Oswestry disability score (ODI); The decrease in irradiation received will be collected, compared to that of the conventional fluoroscopic technique.

DETAILED DESCRIPTION:
Foraminal periradicular infiltrations for therapeutic purposes are currently recognized as an integral part of the treatment of radiculalgia, particularly in case of radiculalgia refractory to a well-conducted initial treatment, in combination with the rehabilitation and education of the patient. The incidence of low back pain, lumbar pain or pure radiculalgia in the general population is very high. In fact, the majority of people will experience at least once in their life low back pain or neck pain, favored by the growing aging of the population. This leads us to propose infiltrative techniques more and more modern, as much in the technique performed as in the type of medication used, presenting the best risk / benefit ratio. Infiltrations guided by imaging tend to become less and less "invasive", with the undeniable contribution of ultrasound as a major tool in the diagnostic and therapeutic approaches, both in specialized pain management clinic as in other medical specialties. To date, infiltrations are still mostly performed under fluoroscopic control by injection of contrast medium (epidurography), or under CT control, where the identification of the anatomical structures and therefore the target allows a greater accuracy of the level of infiltration. These two techniques have proven their effectiveness, but have significant disadvantages, such as the irradiation of the patient as well as that of the practitioner because of the number of daily acts performed; their cost, and the need for a radiologist in the case of a CT technique. For its part, ultrasound is easily available, easy to use, represents a lower cost, and the lack of irradiation.

In recent years ultrasound has proved effective in identifying anatomical structures of the spine and in the techniques of lumbar periradicular infiltration, whether performed in sagittal paramedian or oblique sagittal paramedian, the latter having shown a better intra-foraminal distribution of the injected product. (39.5% vs 87.5% in terms of intraforaminal diffusion of the contrast medium). In addition, teams have shown the superiority of ultrasound-guided lumbar foraminal infiltration compared with CT control in terms of time spent on infiltration, for exact accuracy in 90% of patients, and an improvement in radiculalgia at 1 month similar between the two techniques.

We propose here to evaluate the precision of lumbar periradicular infiltration performed under a transverse ultrasound approach by performing a fluoroscopic control once the needle in the desired position. The effectiveness of the technique will be assessed by measuring different pain and disability scores at four weeks post-infiltration: the Visual analogue pain scale score, the DN4 score, and the Oswestry disability score (ODI); The decrease in irradiation received will be collected, compared to that of the conventional fluoroscopic technique.

ELIGIBILITY:
Inclusion Criteria:

* neurology, neurosurgery, physical medicine, algology consultation
* over the age of 18
* Radiculalgia in the territory corresponding to the root lesion
* Symptomatology inferior to two months.
* Imaging (CT scan or MRI) or electromyographic study with evidence (foraminal disc herniation or foraminal stenosis) of the irritation or the causal compression of the radicular symptomatology

Exclusion Criteria:

* allergy to any of the constituents of the infiltrated product, or to the contrast medium
* unstable medical condition: cardiac, respiratory, endocrine (uncontrolled diabetes)
* inability to put himself in a prone position
* depression: HADS score equal to or greater than 11.
* root lesion caused by an accident at work, a tumoral or infectious causal process.
* local infection (cutaneous, perimedullary / spinal) or systemic
* coagulopathy (platelets <50000 / mm3, Prothrombin time <60%, INTernational normalized ratio> 1.5), anticoagulant or antiplatelet therapy treatment other than aspirin
* Lumbar surgical history
* history of foraminal or perimedullary infiltration of less than 6 months
* symptoms older than two months
* pregnant woman

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-02-27 (Actual); Primary Completion 2018-04-30 (Estimated); Study Completion 2018-05-30 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of needle placement under ultrasound guidance | Before infiltration
  Good position: G. Wrong position: W.

SECONDARY OUTCOMES:
Irradiation doses | 24h
  centiGray. Radioscopy irradiation doses will be calculated in each procedure, to determine how efficient the ultrasound approach is, compared to fluoroscopy only.
Visual analogue scale | Baseline, 2weeks, 4weeks
  0/10 (minimum) to 10/10 (maximum)
Neuropathic pain score: DN4 | Baseline, 2 weeks, 4 weeks
  Score /10
Oswestry Disability index | Baseline, 2 weeks, 4 weeks
  % out of 50 questions (0/50= 0% to 50/50=100%)

CONTACTS AND LOCATIONS:
Overall Officials: Van Obbergh, Study Director — Chief of staff Anesthesiology
Locations (1):
- Hopital Erasme, Anderlecht, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gangi A, Dietemann JL, Mortazavi R, Pfleger D, Kauff C, Roy C. CT-guided interventional procedures for pain management in the lumbosacral spine. Radiographics. 1998 May-Jun;18(3):621-33. doi: 10.1148/radiographics.18.3.9599387.
- [Result] Galiano K, Obwegeser AA, Bodner G, Freund M, Maurer H, Kamelger FS, Schatzer R, Ploner F. Real-time sonographic imaging for periradicular injections in the lumbar spine: a sonographic anatomic study of a new technique. J Ultrasound Med. 2005 Jan;24(1):33-8. doi: 10.7863/jum.2005.24.1.33. PMID 15615926
- [Result] Obernauer J, Galiano K, Gruber H, Bale R, Obwegeser AA, Schatzer R, Loizides A. Ultrasound-guided versus computed tomography-controlled periradicular injections in the middle and lower cervical spine: a prospective randomized clinical trial. Eur Spine J. 2013 Nov;22(11):2532-7. doi: 10.1007/s00586-013-2916-0. Epub 2013 Jul 23. PMID 23877110
- [Result] Gofeld M, Bristow SJ, Chiu SC, McQueen CK, Bollag L. Ultrasound-guided lumbar transforaminal injections: feasibility and validation study. Spine (Phila Pa 1976). 2012 Apr 20;37(9):808-12. doi: 10.1097/BRS.0b013e3182340096. PMID 21912311
- [Result] Kim YH, Park HJ, Moon DE. Ultrasound-guided Pararadicular Injection in the Lumbar Spine: A Comparative Study of the Paramedian Sagittal and Paramedian Sagittal Oblique Approaches. Pain Pract. 2015 Nov;15(8):693-700. doi: 10.1111/papr.12249. Epub 2014 Oct 14. PMID 25313534